CLINICAL TRIAL: NCT06825169
Title: A Phase I/II, Open Label, Single Arm, Dose Escalation and Dose Expansion Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of Human Induced Pluripotent Stem Cell Derived Mesenchymal Stromal Cells (NCR101) Injection in the Treatment of Subjects With Interstitial Lung Disease
Brief Title: A Trial to Evaluate the Safety, Tolerability and Preliminary Efficacy of NCR101 in the Treatment of Subjects With Interstitial Lung Disease
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nuwacell Biotechnologies Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCR101-1001
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Interstitial Lung Disease (ILD)
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NCR101 injection (Experimental): Cohort1:Low dose NCR101 injection; Cohort2:High dose NCR101 injection
  Interventions: Biological: NCR101 injection

INTERVENTIONS:
Biological: NCR101 injection — Subjects will receive one NCR101 injection in Single Ascending Dose（SAD）and receive 4 NCR101 injections in Multiple Ascending Dose(SAD).

SUMMARY:
The target of this trial is to evaluate the safety, tolerability and preliminary efficacy of NCR101 in the treatment of subjects with interstitial lung disease. The trial contains Single ascending dose（SAD） and Multiple ascending dose（MAD）. Subjects will receive at least 1 dose of NCR101.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) is a group of heterogeneous diseases, including idiopathic pulmonary fibrosis(IPF), hypersensitivity pneumonia, sarcoidosis, and connective tissue-associated interstitial lung disease (CTD-ILD), which is characterized by alveolar unit inflammation and/or fibrinization, leading to the destruction of lung structure and loss of function. In the absence of effective treatment, most ILD may develop diffuse pulmonary fibrosis, leading to structural destruction of lung tissue, diffusion dysfunction, and progressive respiratory failure and death. ILD causes a heavy disease and socio-economic burden, and has become a major public health problem. The target of treatment for interstitial lung disease depends on the type of disease and its clinical manifestations. At present, the existing drugs and treatments such as Pirfenidone and Nintedanib can only alleviate the symptoms of IPF or delay the progression of the disease, and the survival improvement is not obvious, and there is no treatment on the market can cure IPF, Patients with connective tissue have a high burden of lung complications, are prone to ILD complications, and the diagnosis and treatment of ILD are difficult for different CTDs. The evidence to guide the optimization of treatment is limited. Therefore, novel drugs with great therapeutic potential are urgently needed for ILD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old (including threshold), gender not limited;
* Meets the diagnosis of interstitial lung disease;
* Screening for interstitial lung disease diagnosed by pulmonary imaging within the first 6 months;
* For patients undergoing glucocorticoid therapy at the time of screening: the background treatment remained stable during the study period;
* If the patient is undergoing anti-fibrotic therapy (pirfenidone or nintedanib) at the time of screening, they must have received a stable dose for at least 4 weeks at the time of screening and plan to continue receiving this background therapy steadily after entering this study;
* Patients of childbearing age (male and female) must agree to take effective non pharmacological contraceptive measures during the trial period and within 6 months after the last use of medication:
* Voluntarily sign an informed consent form and be able to cooperate in completing research related procedures and checks.

Exclusion Criteria:

* Individuals with a history of severe allergies or allergies to the main active ingredients or excipients of the investigational drug;
* Individuals who have been hospitalized for three or more times due to acute exacerbation of ILD or other respiratory diseases within the previous year prior to screening;
* Individuals with a history of mechanical ventilation (invasive or non-invasive) within the past month prior to screening, or those currently requiring oxygen therapy (oxygen therapy duration>15 hours/day);
* Individuals who have contracted infectious pneumonia or require intravenous anti-infective treatment within the previous month; Previous history of tuberculosis
* Patients with other serious respiratory diseases, such as asthma, those with airway obstruction (FEV1/FVC<0.7 before using bronchodilators), and those with other clinically significant abnormalities in the lungs;
* Within the first 3 days of enrollment, use high-dose corticosteroids (equivalent to methylprednisolone>240 mg/day) or irregularly use systemic corticosteroids;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Event(AE) or Serious Adverse Event(SAE) | 4 weeks after administration of SAD and multiple ascending dose (MAD)
  Number of participants with treatment-related adverse events or serious adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Diffusion capacity of the lungs for carbon monoxide(DLCO) | 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Change from baseline in the result of DLCO
Forced vital capacity (FVC) | 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Change from baseline in the result of FVC
Forced expiratory volume in 1 second (FEV1) | 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Change from baseline in the result of FEV1
6-min walk test (6MWT) | 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Change from baseline in the result of 6MWT
St George's Respiratory Questionnaire (SGRQ) | 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Change from baseline in the result of SGRQ
Dyspnea index | 4 weeks, 12 weeks, 24 weeks, 48 weeks
  Change from baseline in the result of Dyspnea index
high-resolution computed tomography (HRCT) Score | 24 weeks, 48 weeks
  Change from baseline in the result of

CONTACTS AND LOCATIONS:
Overall Officials: Tao Ren, MD, Principal Investigator — Shanghai 6th People's Hospital